CLINICAL TRIAL: NCT03184077
Title: Rapidly Absorbing Polyglactin 910 Versus Poliglecaprone 25 for Laceration Repair: A Randomized Controlled Trial
Brief Title: Rapidly Absorbing Polyglactin 910 Versus Poliglecaprone 25 for Laceration Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20000992
Record Dates: First submitted 2017-04-19; First posted 2017-06-12 (Actual); Results first posted 2018-08-08 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Dyspareunia; Perineal Tear; Sutured Laceration
Keywords: Postpartum dyspareunia; Obestric laceration
MeSH Terms: conditions — Dyspareunia | interventions — Polyglactin 910; glycolide E-caprolactone copolymer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Polyglactin 910 (Active Comparator)
  Interventions: Procedure: Laceration Repair with Polyglactin 910
- poliglecaprone 25 (Active Comparator)
  Interventions: Procedure: Laceration Repair with poliglecaprone 25

INTERVENTIONS:
Procedure: Laceration Repair with Polyglactin 910 — Polyglactin 910 suture for laceration repair
  Arms: Polyglactin 910
Procedure: Laceration Repair with poliglecaprone 25 — poliglecaprone 25 suture for laceration repair
  Arms: poliglecaprone 25

SUMMARY:
To evaluate the rates of dyspareunia with rapidly absorbing polyglactin 910 compared to poliglecaprone 25 using a validated sexual function questionnaire.

To assess maternal satisfaction with the laceration repair and suture material.

To assess overall perineal pain using a visual analog scale.

To assess the rate of wound breakdown and the need for suture removal.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted and VCU medical center comparing 2 types of suture: rapidly absorbing polyglactin 910 (Vicryl Rapide) and poliglecaprone 25 (Monocryl) for first and second-degree lacerations requiring suture repair. Patients will be enrolled in the study immediately after vaginal delivery if a laceration occurs spontaneously. Patients will be randomized to one of the 2 sutures after enrollment.

Randomization will be obtained via computer generation in consecutively numbered, opaque sealed envelopes with the name of one of the suture materials. The envelope will be opened at the time of repair of perineal laceration once inclusion criteria have been met by the physician or midwife performing the laceration repair. Repair with the chosen suture will be performed using the continuous suture technique using a 3-0 suture, which is current standard practice. Patients will not be informed of the type of suture used, although the type of suture will be recorded in the patient's electronic medical record. Various maternal and fetal characteristics will be recorded including maternal age, gravity and parity, gestational age at delivery, birth weight, mode of vaginal delivery (spontaneous or operative).

Pain will be evaluated using a numeric pain scale at their 6 week postpartum visit and at 3 months postpartum via a telephone interview. At 3 months postpartum they will also be asked the following questions - Have you resumed sexual intercourse(yes/no)? How long after delivery was it before you resumed intercourse? Did you have pain the first time after delivery (yes/no)? Do you have continued dyspareunia (1-10)? Do you have residual perineal pain unrelated to intercourse? How satisfied are you with your laceration repair (very unsatisfied -1, neutral-3, very satisfied- 5). They will also be administered a 6 question validated Female Sexual Function Index.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, patients with first and second degree spontaneous lacerations or those with midline or mediolateral epsiotomies that were uncomplicated, and hemodynamically stable paitents

Exclusion Criteria:

* non-english speaking, women without laceration or with more extensive third or fourth degree lacerations, and inmates

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 318 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2017-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley W Carroll, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyglactic 910 (Vicryl Rapide): Laceration Repair with Polyglactic 910 (Vicryl Rapide): Polyglactic 910 suture for laceration repair
- Monocryl: Laceration Repair with Monocryl: Monocryl suture for laceration repair
Period: Overall Study
Arm/Group | Polyglactic 910 (Vicryl Rapide) | Monocryl
Started | 166 | 152
Completed | 145 | 131
Not Completed | 21 | 21
Not completed — Lost to Follow-up | 21 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyglactic 910 (Vicryl Rapide) | Monocryl | Total
Number analyzed (Participants) | 145 | 131 | 276
Age, Continuous [Mean (Full Range); unit: years] | 27.4 [19 to 42] | 27.6 [18 to 40] | 27.4 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 131 | 276
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 63 | 51 | 114
  White | 60 | 62 | 122
  Asian | 4 | 5 | 9
  Hispanic or Latino | 6 | 1 | 7
  Other | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 145 | 131 | 318

OUTCOME MEASURES:

1. Primary Outcome: Rates of Dyspareunia
Description: To evaluate the rates of dyspareunia with rapidly absorbing polyglactin 910 compared to poliglecaprone 25 using a validated sexual function questionnaire, with higher scores indicating greater discomfort or pain.
  Scale used - Female Sexual Function Index -6 where 0 indicates no sexual activity, 1 indicates a worse outcome and 5 indicates a better outcome.
  The scale assesses sexual desire, arousal, lubrication, orgasm, sexual satisfaction and sexual pain.
  A score of 1 indicates very low desire, arousal, almost never or never becoming lubricated or achieving orgasm, being very dissatisfied with sexual life and almost always or always having pain with intercourse.
  A score of 5 indicates very high desire, arousal, almost always or always becoming lubricated or achieving orgasm, being very satisfied with sexual life and almost never or never having pain with intercourse.
Time Frame: 3 months postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Polyglactin 910 (Vicryl Rapide): Laceration Repair with Polyglactin 910 (Vicryl Rapide): Polyglactin 910 suture for laceration repair
Arm/Group | Polyglactin 910 (Vicryl Rapide) | Poliglecaprone 25
Number analyzed (Participants) | 145 | 131
units on a scale | 3.6 (1.4) | 3.49 (1.47)
Statistical Analysis 1: Comparison: Polyglactin 910 (Vicryl Rapide) vs Poliglecaprone 25; Test type: Superiority; p = 0.16, Chi-squared

2. Secondary Outcome: Postpartum Pain
Description: To assess overall perineal pain using a visual analog scale on a range of 0-10, with 0 being no pain and 10 being worst imaginable pain Scale used - Pain Numeric Rating Scale. A minimal score of 0 indicates no pain whereas a maximums core of 10 indicates the worse imaginable pain.
Time Frame: 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polyglactin 910 (Vicryl Rapide) | Poliglecaprone 25
Number analyzed (Participants) | 145 | 131
units on a scale | .85 (1.67) | .83 (1.62)
Statistical Analysis 1: Comparison: Polyglactin 910 (Vicryl Rapide) vs Poliglecaprone 25; Test type: Superiority; p = 0.62, Chi-squared

3. Secondary Outcome: Overall Sexual Function
Description: Level of sexual desire or interest on a scale of 1-5, with 5 being the highest level of interest
  Scale used - Female Sexual Function Index -6 where 0 indicates no sexual activity, 1 indicates a worse outcome and 5 indicates a better outcome.
  The scale assesses sexual desire, arousal, lubrication, orgasm, sexual satisfaction and sexual pain.
  A score of 1 indicates very low desire, arousal, almost never or never becoming lubricated or achieving orgasm, being very dissatisfied with sexual life and almost always or always having pain with intercourse.
  A score of 5 indicates very high desire, arousal, almost always or always becoming lubricated or achieving orgasm, being very satisfied with sexual life and almost never or never having pain with intercourse.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polyglactin 910 (Vicryl Rapide) | Poliglecaprone 25
Number analyzed (Participants) | 145 | 131
units on a scale | 2.87 (1.4) | 2.51 (1.47)
Statistical Analysis 1: Comparison: Polyglactin 910 (Vicryl Rapide) vs Poliglecaprone 25; Test type: Superiority; p = 0.01, Chi-squared — This is a calculated p value

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Polyglactic 910 (Vicryl Rapide) | Monocryl
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/152
Other Adverse Events (participants affected / at risk) | 0/166 | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT03184077/Prot_SAP_000.pdf